CLINICAL TRIAL: NCT00545376
Title: The Use of Osteopathic Manipulation in a Clinic and Home Setting to Address Pulmonary Distress as Related to Asthma in Southwest Virginia
Brief Title: Effect of OMT on Asthma Symptoms in Southwest Virginia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edward Via Virginia College of Osteopathic Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F-12
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Manipulation, Osteopathic; Ambulatory Care Facilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (No Intervention): This group will leave after the first visit without additional instruction and will be asked to return in two weeks for a follow up lung assessment.
- 2 (Experimental): This group, at the first visit, will be taught three home OMT techniques that a family member or friend can administer to them. They will be asked to do these techniques at least 4 times a week, up to every day, for two weeks before returning for a follow up lung assessment.
  Interventions: Procedure: Osteopathic Manipulative Treatment - in clinic; Procedure: Osteopathic Manipulative Treatment - at home
- 3 (Experimental): This arm is the physicians that I will recruit participants through. They will be exposed to education about the use of OMT for asthma.
  Interventions: Other: Education to physicians

INTERVENTIONS:
Procedure: Osteopathic Manipulative Treatment - in clinic — I will do a thoracic/rib screening and treatment with muscle energy or facilitated positional release, a diaphragm soft tissue release, suboccipital release, and a thoracic compression. This treatment takes 10 minutes and is only done at the first visit.
  Arms: 2
Procedure: Osteopathic Manipulative Treatment - at home — One group will learn how to do three home OMT techniques: suboccipital release, pectoral traction, and rib raising. They will be asked to do this at least 4 times a week for two weeks.
  Arms: 2
Other: Education to physicians — I will educate physicians using demonstration and reading material as to the possible benefits of incorporating it into the treatment of asthma.
  Arms: 3

SUMMARY:
There is a high prevalence of asthma in southwest Virginia and there are multiple osteopathic manipulative techniques (OMT) which are thought to improve lung function. However, there are inadequate studies regarding the effectiveness of using osteopathic manipulative treatment (OMT) as an office treatment or a home treatment to address obstructive lung disease. In addition, there is little information on the level of acceptance, use, and cost effectiveness of using OMT in rural southwest Virginia. The purpose of this study is to determine the viability of OMT treatment with asthma, the level of acceptance in selected clinics in southwest Virginia, and the effectiveness of home OMT education in order to implement a program to improve asthma control. The study hypotheses are: 1. Osteopathic manipulation delivered to the asthmatic patient will significantly improve spirometry values, thoracic excursion, and subjective asthma symptoms. (.05 alpha) 2.Patients who are taught and use a home treatment regime for asthma will significantly improve spirometry values, thoracic excursion, and subjective asthma symptoms after two weeks, compare with those who do not have home treatment.

3.Physicians educated on the use of OMT for asthma will increase their perceived future use of OMT as an adjunct to treat this disorder.

DETAILED DESCRIPTION:
In this study, participants will be recruited from several family practice, pulmonologist, and asthma specialist offices in southwest Virginia. These participants will undergo two visits. At the first visit, a lung assessment comprised of three components will be performed, then a 10 minute OMT session, then the lung assessment will be repeated. The lung assessment includes a patient symptom survey, a thoracic excursion measurement, and spirometry. The participants will then be divided into one of two groups. Group 1 will have no further instruction while group 2 will be taught some simple home OMT techniques and asked to do them at home. Both groups will return two weeks later for a follow up lung assessment. Results when then be studied to determine the effect of OMT on lung function in asthmatics as well as the effect of incorporating home OMT. In addition, physicians will be involved in learning about OMT and these techniques and they will be assessed for a change in attitude, awareness, and willingness to incorporate OMT when applicable.

ELIGIBILITY:
Inclusion Criteria:

* Age 5-55
* mild intermittent, mild persistent, or moderate persistent asthma

Exclusion Criteria:

* severe persistent asthma
* congestive heart failure
* active pulmonary infection
* oral steroid burst in past month
* hospitalization for pulmonary causes in past three months
* OMT treatment directed towards thoracic and ribs in past three months

Ages: 5 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2007-10; Primary Completion 2008-01 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Mini-AQLQ | 2 weeks
patient symptoms | pre and post OMT and follow-up
thoracic excursion | pre and post OMT and follow up
spirometry | pre and post OMT and follow up

SECONDARY OUTCOMES:
physician acceptance survey | pre and post study

CONTACTS AND LOCATIONS:
Overall Officials: Macy L Latter, Principal Investigator — VCOM
Locations (1):
- VCOM, Blacksburg, Virginia, United States